CLINICAL TRIAL: NCT07405918
Title: 3D Printed Customized Bone Graft for Alveolar Regeneration: Longitudinal Cohort Evaluation
Status: Not yet recruiting | Type: Observational
Sponsor: University of Guarulhos (Other)
Responsible Party: Principal Investigator, Jamil awad shibli, Principal Investigator, University of Guarulhos
Other Study IDs: Guaruhos University
Record Dates: First submitted 2026-01-21; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Periodontal Diseases; Periodontal Bone Loss
Keywords: Personalized bone graft; 3D printed customized bone block; Guided Bone Regeneration; Personalized Medicine
MeSH Terms: conditions — Periodontal Diseases; Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical evaluation — Clinical parmeters and radiographical analysis

SUMMARY:
This study will evaluate the behavior of the implant-supported restorations (prosthesis) placed into the areas grafted with the 3D printed customized bone (personalized graft produced to fit a specific bone defect), as well as the volume contraction of the printed bone.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* over 18 years of age
* Subjects that received regenerative surgical treatment by customized 3D printed blocks.
* Subjects must agree to participate in the study and agree to sign the Informed Consent.

Exclusion Criteria:

* Subjects with ilness that avoid their presence to the clinical evaluation
* ISubjects who have lost the customized blocks
* Subjects who do not agree to participate in the study will be excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This prospective cohort study will evaluate the peri-implant conditions of patients who received regenerative procedures using 3D-printed blocks at the UnG Clinic. To this end, participants will be selected from the UnG graduate clinic who received the regenerative treatment using 3D-printed blocks between 2019 and 2025. Participants selected for the study must sign the Informed Consent Form (ICF) after a verbal and written explanation of the project. Subjects will receive oral hygiene instruction and professional prophylaxis prior to clinical examinations.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal Clinical Parameter of the implants Placed in the Grafted area | 5 years
  Marginal Bone Loss < 2mm

SECONDARY OUTCOMES:
Bone Graft Volume Alteration | 6 years
  Tomographic Volumetric Measurement (mm3) of the 3D printed graft after a period ranged between 1 to 6 years

IPD SHARING:
Plan to Share IPD: Undecided